CLINICAL TRIAL: NCT05673577
Title: A Phase II Study of Camrelizumab in Combination With Cetuximab and Chemotherapy as First-line Therapy for Patients With Relapsed/Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: Camrelizumab in Combination With Cetuximab and Chemotherapy for Relapsed/Metastatic HNSCC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-HN-001
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Chemo-naive HNSCC; PD-1 inhibitor; cetuximab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+cetuximab+chemotherapy (Experimental): Camrelizumab: 200mg vgtt q3w, 3 weeks as a cycle; Cetuximab first dose 400mg/m2, vgtt, following by 250 mg/m2 after first dose, qw, 3 weeks as a cycle; albumin paclitaxel: 125mg/m2, vgtt, d1, 8, q3w，for up to 6 cycles; cisplatin: 75mg/m2, vgtt，d1，q3w, for up to 6 cycles;
  Then, in maintenance therapy, Camrelizumab: 200mg vgtt q2w; Cetuximab 500mg/m2, vgtt q2w until intolerable toxicity or disease progression
  Interventions: Drug: Camrelizumab+cetuximab+chemotherapy

INTERVENTIONS:
Drug: Camrelizumab+cetuximab+chemotherapy — Camrelizumab: 200mg vgtt q3w, 3 weeks as a cycle; Cetuximab first dose 400mg/m2, vgtt, following by 250 mg/m2 after first dose, qw, 3 weeks as a cycle; albumin paclitaxel: 125mg/m2, vgtt, d1, 8, q3w，for up to 6 cycles; cisplatin: 75mg/m2, vgtt，d1，q3w, for up to 6 cycles;
  Then, in maintenance therapy, Camrelizumab: 200mg vgtt q2w; Cetuximab 500mg/m2, vgtt q2w until intolerable toxicity or disease progression

SUMMARY:
This is a single-center, single-arm, phase 2 study to evaluate the efficacy and safety of camrelizumab in combination with cetuximab and chemotherapy as first-line for patients with relapsed/metastastic head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
Patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) not amenable to curative-intent therapies have poor survival.

At present, the standard treatment is cetuximab and chemotherapy plus PD-1 inhibitor Regimen.

This study is a phase II, prospective, single arm，single-center study, which requires a total of 40 R/M HNSCC patients. Patients will receive no more than 6 cycles of albumin paclitaxel and cisplatin, repeated every 3 weeks. PD-1 inhibitor will be administered until progression every 3 weeks. Cetuximab will be administered 400 mg/m2 at first dose, following by 250 mg/m2 after first dose until progression, repeated every 3 weeks.

ELIGIBILITY:
Main inclusion Criteria:

1. Histologically- or cytologically-confirmed recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) HNSCC.
2. Patients with distant metastases, or patients with local recurrence who are not suitable for local radical therapy, must have previously received radiotherapy (postoperative radiotherapy or radical radiotherapy) for local recurrence and must have ended radiotherapy more than 6 months ago.
3. Patients who have not received systemic chemotherapy before and who have received systemic chemotherapy as part of multidisciplinary treatment 6 months ago for locally advanced disease can be enrolled.
4. Age 18-70 years old.
5. ECOG performance status 0-1.
6. Patients must have at least one lesion that can be evaluated by enhanced CT or MRI according to Recist v1.1.
7. Hematopoietic function of bone marrow is basically normal: WBC ≥ 3.5 × 109/L, ANC ≥ 1.5 × 109/L, PLT ≥ 80 × 109/L, Hb ≥ 90 g/L.
8. Liver and kidney functions are basically normal: total bilirubin, ALT and AST are all<1.5 × UNL (upper limit of normal value); Cr < 1.5 × UNL, and creatinine clearance ≥ 50 ml/min.
9. Patients must have a life expectancy of at least 3 months.
10. Patients volunteered to sign informed consent.

Main exclusion Criteria:

1. Patients with a known history of severe allergy to monoclonal antibody therapy.
2. Patients with previous camrelizumab therapy or previous cetuximab therapy (cetuximab as part of therapy in multidisciplinary therapy for curative purposes may be included).
3. Patients with clinically significant heart disease, including severe cardiac insufficiency: New York College of Cardiology (NYHA) Grade IV cardiac insufficiency, unstable angina, acute myocardial infarction within 6 months prior to screening, congestive heart failure, Q-Tc interval greater than 500ms.
4. Patients who had received secondary or higher gardes surgery within 3 weeks prior to treatment.
5. Patients suffering from autoimmune disease requiring treatment, or syndrome history requiring systemic use of steroids/immunosuppressants, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.
6. Other serious and uncontrollable concomitant diseases that may affect the compliance of the scheme or interfere with the interpretation of the results, including uncontrollable diabetes, or pulmonary diseases (interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm history).
7. Patients have evidence of central nervous system disease.
8. Patients with known hepatitis B (HBV) (HBsAg positive and HBV DNA ≥ 103IU/ml) and hepatitis C (HCV) infection (HCV antibody positive and HCV RNA detectable); And other subjects with acquired and congenital immunodeficiency diseases, including but not limited to those infected with AIDS virus.
9. Pregnant or lactating woman.
10. Patients have serious active infection.
11. Patients have a history of serious neurological or psychiatric diseases, including dementia or epilepsy.
12. Patients may interfere with the drug abuse, medical, psychological or social conditions of the subject involved in the study or the evaluation of the study results.
13. Patients considered unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years after enrollment of final patient
  Objective response rate measured as number of complete and partial response divided by the number of patients included.

SECONDARY OUTCOMES:
Adverse events | Since the signing of informed consent forms to 30 days after the last cycle
  Hematologic and non hematologic adverse event (CTCAE 5.0）
Progression-free Survival (PFS) | up to 2 years
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival (OS) | up to 2 years
  Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No